CLINICAL TRIAL: NCT00501657
Title: Effects of Sitagliptin on Gastric Emptying in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Royal Adelaide Hospital (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Karen Jones, Professor, Royal Adelaide Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 061025
Record Dates: First submitted 2007-07-13; First posted 2007-07-16 (Estimated); Last update posted 2015-10-29 (Estimated); Status verified 2014-12

CONDITIONS: Gastroparesis; Diabetes Mellitus
Keywords: gastric emptying; glycemia; appetite; incretin hormones
MeSH Terms: conditions — Gastroparesis; Diabetes Mellitus | interventions — Sitagliptin Phosphate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sitagliptin (100mg) (Experimental): Active drug (sitagliptin)
  Interventions: Drug: Sitagliptin
- Placebo (sugar pill) (Placebo Comparator): Inactive drug (placebo)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sitagliptin — 100mg mane for 2 days
  Other Names: MK-0431-075; Januvia
  Arms: Sitagliptin (100mg)
Drug: Placebo — 100mg mane for 2 days
  Arms: Placebo (sugar pill)

SUMMARY:
The purpose of this study is to determine the effects of the drug, sitagliptin, on the rate at which the stomach empties, and the release of gut hormones and blood glucose concentrations, after a mashed potato meal in healthy subjects. Sitagliptin has been shown to reduce the blood glucose (sugar) response to a meal and this may potentially be due to slowing of stomach emptying. This is particularly relevant to people who have diabetes, in whom normalization of elevated blood glucose levels is important to maintain health.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the effect of sitagliptin on gastric emptying, intragastric meal distribution, postprandial glycemia and insulinemia in healthy subjects. Glucagon-like peptide-1 (GLP-1) inhibits gastric emptying, thereby slowing the delivery of nutrients, and their absorption, across the small intestine. The rate of entry of carbohydrate into the small intestine is especially important in patients with diabetes mellitus. Sitagliptin is an orally administered inhibitor of dipeptidyl-peptidase-IV (DPP-IV), the enzyme responsible for the degradation of GLP-1. It is hypothesized that sitagliptin will increase the GLP-1 response to, and thereby slow gastric emptying and diminish the glycemic response to, a carbohydrate-containing meal.

Fifteen healthy subjects (male and female) will be studied. Each subject will be studied on two occasions following treatment for 2 days with sitagliptin (100mg once daily) or matching placebo in a randomized, double blind, crossover design. Measurements of gastric emptying, intragastric meal distribution, blood glucose concentrations, gut hormones and appetite will be measured for 4 hours following ingestion of a mashed potato meal.

ELIGIBILITY:
Inclusion Criteria:

* Male or female (females must be using an appropriate contraceptive method)
* 18 - 45 years
* Body mass index (BMI) 19 - 25 kg/m2.

Exclusion criteria:

* Subjects with gastrointestinal disease, history of gastrointestinal surgery and/or significant gastrointestinal symptoms
* Subjects taking medication known to influence gastrointestinal function
* Alcohol intake > 20 g per day
* Smoking > 10 cigarettes per day
* Pregnant and/or lactating females
* Calculated creatinine clearance < 60 ml/min
* Exposure to ionising radiation for research purposes in the previous 12 months.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2007-07; Primary Completion 2008-06 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Gastric emptying rate | 4 hours per study

SECONDARY OUTCOMES:
Intragastric distribution, gastrointestinal hormone release (GLP-1, GIP), glycemia, insulinemia, appetite | 4 hours per study

CONTACTS AND LOCATIONS:
Overall Officials: Karen L Jones, PhD, Principal Investigator — University of Adelaide, Royal Adelaide Hospital
Locations (1):
- Discipline of Medicine, Royal Adelaide Hospital, Adelaide, South Australia, Australia

REFERENCES:
- [Derived] Stevens JE, Horowitz M, Deacon CF, Nauck M, Rayner CK, Jones KL. The effects of sitagliptin on gastric emptying in healthy humans - a randomised, controlled study. Aliment Pharmacol Ther. 2012 Aug;36(4):379-90. doi: 10.1111/j.1365-2036.2012.05198.x. Epub 2012 Jun 28. PMID 22738299
- See also: Pubmed abstract — http://www.ncbi.nlm.nih.gov/pubmed/22738299